CLINICAL TRIAL: NCT02175095
Title: 3'-Deoxy-3'-18F-fluorothymidine Positron Emission Tomography ([18F] FLT-PET) for the Prediction of Response to Regorafenib in the Metastatic Colorectal Cancer Patients Who Progressed After All Standard Therapies
Brief Title: [18F]FLT-PET as a Predictive Imaging Biomaker of Treatment Responses to Regorafenib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yong Sang Hong, Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLT-PET-regorafenib
Record Dates: First submitted 2014-06-23; First posted 2014-06-26 (Estimated); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer
Keywords: regorafenib; fluorothymidine; positron emission tomography; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Intervention Model Description: This is a imaging biomarker study to evaluate feasibility of [18F]FLT-PET as a potential candidate for predictive imaging biomarker of regorafenib treatment in mCRC patients who progressed after prior standard therapies.
  The mCRC patients who failed to all 3 active cytotoxic chemotherapy (fluoropyrimidines, oxaliplatin and irinotecan) with or without targeted agents will be accrued. Patients will be scheduled to perform [18F]FLT-PET scans before and on 21st day from the administration of regorafenib.
  Regorafenib will be administered 160 mg/day given orally on day 1 to days 21 following 7 days break, which consists of 4 weeks as 1 cycle.
  Standard anatomical response evaluation will be performed every 8 weeks (without regard to the cycles or schedules of chemotherapy). Additional [ 18F]FDG-PET will be performed before treatment and at 21 days after treatment.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib and FLT-PET (Experimental): After checking the eligibility for the study entry, patients will be scheduled to perform [18F]FLT-PET scans before and on 21st day from the administration of regorafenib. Regorafenib will be administered 160 mg/day given orally on day 1 to days 21 following 7 days break, which consists of 4 weeks as 1 cycle. Treatment will be repeated every 4 weeks and continued until disease progression, unacceptable toxicity or the patient's refusal. Standard anatomical response evaluation will be performed every 8 weeks (without regard to the cycles or schedules of chemotherapy). Additional [18F]FDG-PET will be performed before treatment and at 8 weeks (just once at the point of first response evaluation).
  Interventions: Drug: Regorafenib; Diagnostic Test: [18F]FLT-PET; Diagnostic Test: [18F]FDG-PET

INTERVENTIONS:
Drug: Regorafenib — Regorafenib will be administered 160 mg/day given orally on day 1 to days 21 following 7 days break, which consists of 4 weeks as 1 cycle. Treatment will be repeated every 4 weeks and continued until disease progression, unacceptable toxicity or the patient's refusal.
  Other Names: Stivarga
Diagnostic Test: [18F]FLT-PET — [18F]FLT-PET scans before and on 21st day from the administration of regorafenib.
Diagnostic Test: [18F]FDG-PET — [18F]FDG-PET will be performed before treatment and at 21 days after treatment.

SUMMARY:
Regorafenib is approved in the treatment for metastatic colorectal cancer patients who have been progressed after standard therapies, however, there has not been a predictive biomarker. The investigators designed this study to investigate whether [18F]FLT-PET might paly a role as a predictive imaging biomarker of treatment responses to regorafenib.

DETAILED DESCRIPTION:
Recent advances have been made in the treatments for the patients with metastatic colorectal cancer (mCRC) owing to the introductions of targeted agents, which included bevacizumab, cetuximab, panitumumab, and aflibercept. And in addition, regorafenib, a newer tyrosine kinase inhibitor (TKI), has been approved in the treatment for the mCRC patients.

Regorafenib (BAY 73-4506) is an orally available multikinase inhibitor with activity against multiple targets, including tumor angiogenesis (VEGFR-1, -2, -3 and TIE-2), oncogenesis (KIT, RET, RAF-1, BRAF, and BRAFV600E), and tumor microenvironment (PDGF and FGFR). Regorafenib has shown antitumor activities in multiple solid tumors, and demonstrated significant efficacy outcomes in patients with advanced gastrointestinal stromal tumors and colorectal cancers.

The CORRECT study, which compared regorafenib vs placebo in mCRC patients who have been treated with all standard treatment, showed survival improvements with statistical significances; median OS 6.4 vs 5.0 months, HR 0.77, p=0.0052; median PFS 1.9 vs 1.7 months, HR 0.49, p<0.000001. Above these results, regorafenib monotherapy has been recently approved for the treatment of mCRC patients who have been refractory to all of standard therapies.

However, there are still only a few biomarkers which have been established as predictive of treatment responses in the fields of treatments for mCRC patients; KRAS or BRAF mutations for the lack of responses to anti-EGFR agents, cetuximab or panitumumab. There still has not been any biomarker which would be predictive of treatment responses to bevacizumab, aflibercept or regorafenib. The difficulties in search for biomarkers for these agents might come from the facts as following; either bevacizumab or aflibercept does not act directly against tumor itself and should be combined with cytotoxic agents to show efficacy; regorafenib is a multikinase inhibitor which has too many potential targets.

Above these reasons, imaging modalities can be fascinating and alternative candidates for predictive biomarkers of treatment responses. Conventional anatomic imaging studies such as computed tomography (CT) scans can hardly predict the treatment responses earlier, and the RECIST using CT scans, which is widely used for measurement of treatment responses, might have several limitations for measurement of efficacy from targeted agents such as cystic necrosis without tumor shrinkage. In the CORRECT study, overall response rate by RECIST was only 1%, although the rates for disease stabilization was up to 40%, which might be a good example for the limitations of the RECIST using conventional anatomical imaging studies for the response evaluation of regorafenib.

Among imaging studies, PET scans are useful tools for the noninvasive measurement of functional changes after treatment with targeted agents, and [18F]FLT-PET is potentially useful tool for earlier prediction of treatment responses because it can detect earlier changes of cellular proliferation using [18F]FLT (fluorothymidine), a radiotraceable substitute for thymidine which is essential for DNA synthesis. Several studies have been reported that [18F]FLT-PET may allow an early assessment of the response to chemotherapy including targeted agents. There also has been a report that [18F]FLT-PET could predict treatment responses of BRAF inhibitors in the colorectal cancer xenograft model; regorafenib also has an inhibitory effect on BRAF.

Therefore, the investigators have planned this study with hypothesis that [18F]FLT-PET could be useful for identifying a subgroup of mCRC patients with clinical responsiveness to regorafenib.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the colon or the rectum.
2. Progressed after 3 active cytotoxic chemotherapy including fluoropyrimidines, oxaliplatin and irinotecan during or within 6 months of their administrations with or without targeted agents (bevacizumab or cetuximab).
3. Extrahepatic measurable lesion(s) by RECIST 1.1.
4. Unresectable metastatic disease.
5. Age over 20 years old.
6. Have a life expectancy of at least 3 months.
7. ECOG performance status of 1 or lower.
8. Adequate organ functions.
9. Be willing and able to comply with the protocol for the duration of the study.
10. Give written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw the study at any time, without prejudice.
11. Women of childbearing potential and men must agree to use adequate contraception since signing of the IC form until at least 8 weeks after the last study drug administration.

Exclusion Criteria:

1. Prior treatment of regorafenib.
2. Liver-limited metastasis.
3. Inability to perform [18F]FLT and [18F]FDG-PET imaging studies due to physical inability or claustrophobia.
4. Concurrent or previous history of another primary cancer within 3 years prior to randomisation except for curatively treated cervical cancer in situ, non-melanomatous skin cancer, superficial bladder cancer (pTis and pT1) and curatively treated thyroid cancer of any stage. Concurrent, histologically confirmed, unresected thyroid cancer without distant metastasis could be allowed with the agreement of the chief principal investigator.
5. Uncontrolled CNS metastases.
6. Prior radiation therapy would be permitted, but non-radiated evaluable lesions should be present at study entry.
7. Uncontrolled hypertension (>150/90 mmHg) despite of optimal management; anti-hypertensive drugs for BP lowering before study entry would be permitted.
8. Congestive heart failure ≥ New York Heart Association (NYHA) class 2.
9. Unstable angina, new-onset angina within 3 months, or history of myocardial infarction within 6 months before the study entry.
10. Arterial or venous thromboembolism within 6 months.
11. Serious concurrent infections or non-malignant illness.
12. Liver cirrhosis ≥ Child-Pugh class B.
13. Active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
14. Peripheral neuropathy of grade ≥ 2.
15. Major surgery or significant traumatic injury within 28 days prior to study treatment.
16. Non-healing wound, ulcer, or bone fracture.
17. Current evidence of significant gastrointestinal bleeding or (impending) obstruction.
18. Any hemorrhage or bleeding event of grade ≥ 3 within 4 weeks prior to the start of study medication.
19. Proteinuria ≥ 3+ in the routine urinalysis; in this case, the total protein in the 24-hour urine collection should be measured, and the accrual is permitted if total protein < 3.5 g/day.
20. Pregnant of breast-feeding subjects. Women of child-bearing potential must have pregnancy test within 7 days and a negative result must be documented before start of study treatment.
21. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
22. Use of strong CYP3A4 inducers or inhibitors which are known to decrease the metabolism of regorafenib (ketoconazole, rifampin, phenytoin, carbamazepine, phenobarbital).
23. Known hypersensitivity to the study drug or any of its excipients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-07-18 (Actual); Primary Completion 2016-08-10 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Sang Hong, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa, South Korea

REFERENCES:
- [Background] Van Cutsem E, Tabernero J, Lakomy R, Prenen H, Prausova J, Macarulla T, Ruff P, van Hazel GA, Moiseyenko V, Ferry D, McKendrick J, Polikoff J, Tellier A, Castan R, Allegra C. Addition of aflibercept to fluorouracil, leucovorin, and irinotecan improves survival in a phase III randomized trial in patients with metastatic colorectal cancer previously treated with an oxaliplatin-based regimen. J Clin Oncol. 2012 Oct 1;30(28):3499-506. doi: 10.1200/JCO.2012.42.8201. Epub 2012 Sep 4. PMID 22949147
- [Background] Bennouna J, Sastre J, Arnold D, Osterlund P, Greil R, Van Cutsem E, von Moos R, Vieitez JM, Bouche O, Borg C, Steffens CC, Alonso-Orduna V, Schlichting C, Reyes-Rivera I, Bendahmane B, Andre T, Kubicka S; ML18147 Study Investigators. Continuation of bevacizumab after first progression in metastatic colorectal cancer (ML18147): a randomised phase 3 trial. Lancet Oncol. 2013 Jan;14(1):29-37. doi: 10.1016/S1470-2045(12)70477-1. Epub 2012 Nov 16. PMID 23168366
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Saltz LB, Clarke S, Diaz-Rubio E, Scheithauer W, Figer A, Wong R, Koski S, Lichinitser M, Yang TS, Rivera F, Couture F, Sirzen F, Cassidy J. Bevacizumab in combination with oxaliplatin-based chemotherapy as first-line therapy in metastatic colorectal cancer: a randomized phase III study. J Clin Oncol. 2008 Apr 20;26(12):2013-9. doi: 10.1200/JCO.2007.14.9930. PMID 18421054
- [Background] Karapetis CS, Khambata-Ford S, Jonker DJ, O'Callaghan CJ, Tu D, Tebbutt NC, Simes RJ, Chalchal H, Shapiro JD, Robitaille S, Price TJ, Shepherd L, Au HJ, Langer C, Moore MJ, Zalcberg JR. K-ras mutations and benefit from cetuximab in advanced colorectal cancer. N Engl J Med. 2008 Oct 23;359(17):1757-65. doi: 10.1056/NEJMoa0804385. PMID 18946061
- [Background] Van Cutsem E, Kohne CH, Hitre E, Zaluski J, Chang Chien CR, Makhson A, D'Haens G, Pinter T, Lim R, Bodoky G, Roh JK, Folprecht G, Ruff P, Stroh C, Tejpar S, Schlichting M, Nippgen J, Rougier P. Cetuximab and chemotherapy as initial treatment for metastatic colorectal cancer. N Engl J Med. 2009 Apr 2;360(14):1408-17. doi: 10.1056/NEJMoa0805019. PMID 19339720
- [Background] Douillard JY, Siena S, Cassidy J, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Oliner KS, Wolf M, Gansert J. Randomized, phase III trial of panitumumab with infusional fluorouracil, leucovorin, and oxaliplatin (FOLFOX4) versus FOLFOX4 alone as first-line treatment in patients with previously untreated metastatic colorectal cancer: the PRIME study. J Clin Oncol. 2010 Nov 1;28(31):4697-705. doi: 10.1200/JCO.2009.27.4860. Epub 2010 Oct 4. PMID 20921465
- [Background] Peeters M, Price TJ, Cervantes A, Sobrero AF, Ducreux M, Hotko Y, Andre T, Chan E, Lordick F, Punt CJ, Strickland AH, Wilson G, Ciuleanu TE, Roman L, Van Cutsem E, Tzekova V, Collins S, Oliner KS, Rong A, Gansert J. Randomized phase III study of panitumumab with fluorouracil, leucovorin, and irinotecan (FOLFIRI) compared with FOLFIRI alone as second-line treatment in patients with metastatic colorectal cancer. J Clin Oncol. 2010 Nov 1;28(31):4706-13. doi: 10.1200/JCO.2009.27.6055. Epub 2010 Oct 4. PMID 20921462
- [Background] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514
- [Background] Demetri GD, Reichardt P, Kang YK, Blay JY, Rutkowski P, Gelderblom H, Hohenberger P, Leahy M, von Mehren M, Joensuu H, Badalamenti G, Blackstein M, Le Cesne A, Schoffski P, Maki RG, Bauer S, Nguyen BB, Xu J, Nishida T, Chung J, Kappeler C, Kuss I, Laurent D, Casali PG; GRID study investigators. Efficacy and safety of regorafenib for advanced gastrointestinal stromal tumours after failure of imatinib and sunitinib (GRID): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):295-302. doi: 10.1016/S0140-6736(12)61857-1. Epub 2012 Nov 22. PMID 23177515
- [Background] Di Nicolantonio F, Martini M, Molinari F, Sartore-Bianchi A, Arena S, Saletti P, De Dosso S, Mazzucchelli L, Frattini M, Siena S, Bardelli A. Wild-type BRAF is required for response to panitumumab or cetuximab in metastatic colorectal cancer. J Clin Oncol. 2008 Dec 10;26(35):5705-12. doi: 10.1200/JCO.2008.18.0786. Epub 2008 Nov 10. PMID 19001320
- [Background] Lievre A, Bachet JB, Boige V, Cayre A, Le Corre D, Buc E, Ychou M, Bouche O, Landi B, Louvet C, Andre T, Bibeau F, Diebold MD, Rougier P, Ducreux M, Tomasic G, Emile JF, Penault-Llorca F, Laurent-Puig P. KRAS mutations as an independent prognostic factor in patients with advanced colorectal cancer treated with cetuximab. J Clin Oncol. 2008 Jan 20;26(3):374-9. doi: 10.1200/JCO.2007.12.5906. PMID 18202412
- [Background] Cousin S, Taieb S, Penel N. A paradigm shift in tumour response evaluation of targeted therapy: the assessment of novel drugs in exploratory clinical trials. Curr Opin Oncol. 2012 May;24(3):338-44. doi: 10.1097/CCO.0b013e3283528b73. PMID 22418613
- [Background] Milano A, Perri F, Ciarmiello A, Caponigro F. Targeted-therapy and imaging response: a new paradigm for clinical evaluation? Rev Recent Clin Trials. 2011 Sep;6(3):259-65. doi: 10.2174/157488711796575540. PMID 21682675
- [Background] Desar IM, van Herpen CM, van Laarhoven HW, Barentsz JO, Oyen WJ, van der Graaf WT. Beyond RECIST: molecular and functional imaging techniques for evaluation of response to targeted therapy. Cancer Treat Rev. 2009 Jun;35(4):309-21. doi: 10.1016/j.ctrv.2008.12.001. Epub 2009 Jan 10. PMID 19136215
- [Background] Chen W, Delaloye S, Silverman DH, Geist C, Czernin J, Sayre J, Satyamurthy N, Pope W, Lai A, Phelps ME, Cloughesy T. Predicting treatment response of malignant gliomas to bevacizumab and irinotecan by imaging proliferation with [18F] fluorothymidine positron emission tomography: a pilot study. J Clin Oncol. 2007 Oct 20;25(30):4714-21. doi: 10.1200/JCO.2006.10.5825. PMID 17947718
- [Background] Herrmann K, Wieder HA, Buck AK, Schoffel M, Krause BJ, Fend F, Schuster T, Meyer zum Buschenfelde C, Wester HJ, Duyster J, Peschel C, Schwaiger M, Dechow T. Early response assessment using 3'-deoxy-3'-[18F]fluorothymidine-positron emission tomography in high-grade non-Hodgkin's lymphoma. Clin Cancer Res. 2007 Jun 15;13(12):3552-8. doi: 10.1158/1078-0432.CCR-06-3025. PMID 17575218
- [Background] Kahraman D, Scheffler M, Zander T, Nogova L, Lammertsma AA, Boellaard R, Neumaier B, Ullrich RT, Holstein A, Dietlein M, Wolf J, Kobe C. Quantitative analysis of response to treatment with erlotinib in advanced non-small cell lung cancer using 18F-FDG and 3'-deoxy-3'-18F-fluorothymidine PET. J Nucl Med. 2011 Dec;52(12):1871-7. doi: 10.2967/jnumed.111.094458. Epub 2011 Nov 7. PMID 22065872
- [Background] Kim SJ, Lee JS, Im KC, Kim SY, Park SA, Lee SJ, Oh SJ, Lee DS, Moon DH. Kinetic modeling of 3'-deoxy-3'-18F-fluorothymidine for quantitative cell proliferation imaging in subcutaneous tumor models in mice. J Nucl Med. 2008 Dec;49(12):2057-66. doi: 10.2967/jnumed.108.053215. Epub 2008 Nov 7. PMID 18997037
- [Background] McKinley ET, Smith RA, Zhao P, Fu A, Saleh SA, Uddin MI, Washington MK, Coffey RJ, Manning HC. 3'-Deoxy-3'-18F-fluorothymidine PET predicts response to (V600E)BRAF-targeted therapy in preclinical models of colorectal cancer. J Nucl Med. 2013 Mar;54(3):424-30. doi: 10.2967/jnumed.112.108456. Epub 2013 Jan 22. PMID 23341544
- [Background] Nakajo M, Nakajo M, Kajiya Y, Jinguji M, Nishimata N, Shimaoka S, Nihara T, Aridome K, Tanaka S, Fukukura Y, Tani A, Koriyama C. Diagnostic performance of (1)(8)F-fluorothymidine PET/CT for primary colorectal cancer and its lymph node metastasis: comparison with (1)(8)F-fluorodeoxyglucose PET/CT. Eur J Nucl Med Mol Imaging. 2013 Aug;40(8):1223-32. doi: 10.1007/s00259-013-2424-9. Epub 2013 May 8. PMID 23653240
- [Background] Sohn HJ, Yang YJ, Ryu JS, Oh SJ, Im KC, Moon DH, Lee DH, Suh C, Lee JS, Kim SW. [18F]Fluorothymidine positron emission tomography before and 7 days after gefitinib treatment predicts response in patients with advanced adenocarcinoma of the lung. Clin Cancer Res. 2008 Nov 15;14(22):7423-9. doi: 10.1158/1078-0432.CCR-08-0312. PMID 19010859
- [Background] Hong YS, Kim HO, Kim KP, Lee JL, Kim HJ, Lee SJ, Lee SJ, Oh SJ, Kim JS, Ryu JS, Moon DH, Kim TW. 3'-Deoxy-3'-18F-fluorothymidine PET for the early prediction of response to leucovorin, 5-fluorouracil, and oxaliplatin therapy in patients with metastatic colorectal cancer. J Nucl Med. 2013 Aug;54(8):1209-16. doi: 10.2967/jnumed.112.117010. Epub 2013 Jun 26. PMID 23804324
- [Background] Mross K, Frost A, Steinbild S, Hedbom S, Buchert M, Fasol U, Unger C, Kratzschmar J, Heinig R, Boix O, Christensen O. A phase I dose-escalation study of regorafenib (BAY 73-4506), an inhibitor of oncogenic, angiogenic, and stromal kinases, in patients with advanced solid tumors. Clin Cancer Res. 2012 May 1;18(9):2658-67. doi: 10.1158/1078-0432.CCR-11-1900. Epub 2012 Mar 15. PMID 22421192
- [Background] Strumberg D, Scheulen ME, Schultheis B, Richly H, Frost A, Buchert M, Christensen O, Jeffers M, Heinig R, Boix O, Mross K. Regorafenib (BAY 73-4506) in advanced colorectal cancer: a phase I study. Br J Cancer. 2012 May 22;106(11):1722-7. doi: 10.1038/bjc.2012.153. Epub 2012 May 8. PMID 22568966
- [Background] Wilhelm SM, Dumas J, Adnane L, Lynch M, Carter CA, Schutz G, Thierauch KH, Zopf D. Regorafenib (BAY 73-4506): a new oral multikinase inhibitor of angiogenic, stromal and oncogenic receptor tyrosine kinases with potent preclinical antitumor activity. Int J Cancer. 2011 Jul 1;129(1):245-55. doi: 10.1002/ijc.25864. Epub 2011 Apr 22. PMID 21170960
- [Background] George S, Wang Q, Heinrich MC, Corless CL, Zhu M, Butrynski JE, Morgan JA, Wagner AJ, Choy E, Tap WD, Yap JT, Van den Abbeele AD, Manola JB, Solomon SM, Fletcher JA, von Mehren M, Demetri GD. Efficacy and safety of regorafenib in patients with metastatic and/or unresectable GI stromal tumor after failure of imatinib and sunitinib: a multicenter phase II trial. J Clin Oncol. 2012 Jul 1;30(19):2401-7. doi: 10.1200/JCO.2011.39.9394. Epub 2012 May 21. PMID 22614970

RESULTS

PARTICIPANT FLOW:
Groups:
- Regorafenib and FLT-PET: After checking the eligibility for the study entry, patients will be scheduled to perform [18F]FLT-PET scans before and on 21st day from the administration of regorafenib. Regorafenib will be administered 160 mg/day given orally on day 1 to days 21 following 7 days break, which consists of 4 weeks as 1 cycle. Treatment will be repeated every 4 weeks and continued until disease progression, unacceptable toxicity or the patient's refusal. Standard anatomical response evaluation will be performed every 8 weeks (without regard to the cycles or schedules of chemotherapy). Additional [18F]FDG-PET will be performed before treatment and at 8 weeks (just once at the point of first response evaluation).
  Regorafenib: After checking the eligibility for the study entry, patients will be scheduled to perform [18F]FLT-PET scans before and on 21st day from the administration of regorafenib. Regorafenib will be administered 160 mg/day given orally on day 1 to days 21 following 7 days break, which consists of 4 weeks as 1 cycle. Treatment will be repeated every 4 weeks and continued until disease progression, unacceptable toxicity or the patient's refusal. Standard anatomical response evaluation will be performed every 8 weeks (without regard to the cycles or schedules of chemotherapy).
Period: Overall Study
Arm/Group | Regorafenib and FLT-PET
Started | 68
Completed | 65
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Between July 2014 and June 2016, we enrolled 68 patients with mCRC who showed progression after all standard therapies, and initiated Regorafenib administration (160 mg/day) at Asan Medical Center in Seoul, Republic of Korea.
Groups:
- Regorafenib and FLT-PET: Baseline characteristics of patients with metastatic colorectal cancer receiving Regorafenib
Arm/Group | Regorafenib and FLT-PET
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 59
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 58 [26 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 26
Region of Enrollment [Number; unit: participants]
  South Korea | 68
ECOG Performance Status 0-1 [Count of Participants; unit: Participants] — GRADE 0=Fully active, able to carry on all pre-disease performance without restriction GRADE 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants | 68
Primary tumour [Count of Participants; unit: Participants]
  Right colon | 11
  Left colon | 25
  Rectum | 32
Histology [Count of Participants; unit: Participants]
  Well differentiated | 7
  Moderately differentiated | 52
  Poorly differentiated | 6
  Mucinous differentiated | 3
Status [Count of Participants; unit: Participants]
  Initially metastatic | 39
  Recurrence with metastasis | 29
Site of metastasis [Count of Participants; unit: Participants] — Radiologic assessments using RECIST 1.1 which is for accurate comparisons between anatomical imaging and [ 18F]FLT-PET scans. Additional CT or MRI scans are highly recommended at the same day when the baseline [18F]FLT-PET is planned
  Participants
    Liver | 28
    Lung | 57
    Lymph node, abdomen | 29
    Peritoenum/omentum | 11
    Bone | 7
    Ovary | 2
RAS status [Count of Participants; unit: Participants]
  Wild | 34
  Mutant | 31
  Unknown | 3
BRAF status [Count of Participants; unit: Participants]
  Wild | 55
  Mutant | 4
  Unknown | 9
Previous targeted agents [Count of Participants; unit: Participants]
  None | 21
  Any | 47
Previous chemotherapy [Count of Participants; unit: Participants]
  2 lines of chemotherapy | 24
  3 lines of chemotherapy | 21
  ≥4 lines of chemotherapy | 23
Previous targeted agents [Count of Participants; unit: Participants] — Population: This status was for the patient who got previous targeted agents.
  Participants
    number analyzed (Participants) | 47
    Anti-VEGF but not anti-EGFR | 28
    Anti-EGFR but not anti-VEGF | 9
    Anti-VEGF and anti-EGFR | 10

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Early Response by 18F-Fluorodeoxyglucose(18F-FDG) Positron Emission Tomography/Computed Tomography (PET/CT) on Day 21 of Regorafenib Compared With the Response Rate of CT RECIST at 8 Weeks
Description: Response assessment using 18F-FDG PET/CT was based on the PERCIST 1.0. The peak SUV value corrected for lean body mass (SULpeak) was measured from the single hottest tumour at each time point. For a tumour to be measurable at baseline, the SULpeak in the target lesion was greater than or equal to 1.5 times the mean SUL in the 3-cm-diameter spherical volume of interest plus two times its standard deviation of the liver. The percentage of change in SULpeak in the measurable target lesion was computed as follows: 100×(SULpeak day 21-SULpeak baseline)/SULpeak baseline. When a non-target lesion showed different responses from the measurable target lesion, we used the overall response considering both the target and non-target responses as previously described.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) by CT scans at 8 weeks.
Time Frame: Regorafenib was administered orally at a dose of 160 mg/day on days 1 to 21 following a 7-day break, with each cycle lasting 4 weeks. Treatment was repeated every 4 weeks and continued until disease progression, unacceptable toxicity, or patient refusal.
Population: Both 18F-FLT and 18F-FDG PET/CT scans were performed in 64 patients; among the remaining four patients, one withdrew consent and three discontinued Regorafenib treatment during the first cycle because of toxicities. With the exception of three patients who had no follow-up CT (n = 2) or no uptake of 18F-FLT (n = 1), 61 were evaluable for the treatment response on both CT and PET/CT in final.
Measure: Count of Participants; unit: Participants
Groups:
- Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) by CT scans at 8 weeks.
  Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), At least a 20% increase in the sum of diameters of target lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
- PET Response Criteria in Solid Tumours (PERCIST): Response assessment using 18F-FDG PET/CT was based on the PERCIST 1.0.
  The peak SUV value corrected for lean body mass (SULpeak) was measured from the single hottest tumour at each time point.
  The percentage of change in SULpeak in the measurable target lesion was computed as follows:
  100×(SULpeak day 21-SULpeak baseline)/SULpeak baseline. When a non-target lesion showed different responses from the measurable target lesion, we used the overall response considering both the target and non-target responses as previously described.
  Complete metabolic response (CMR)= complete resolution of 18F-FDG uptake within the measurable target lesion/disappearance of all other lesions to background blood pool levels/no new suspicious 18F-FDG avid lesions; Partial metabolic response (PMR)=reduction of a minimum of 30% in target measurable tumor 18F-FDG SUL peak, with absolute drop in SUL of at least 0.8 SUL units/no increase >30% of SUL or size in all other lesions; Stable metabolic disease (SMD)=no CMR, PMR, or progressive metabolic disease (PMD); Progressive metabolic disease (PMD)=>30% increase in 18F-FDG SUL peak, with >0.8 SUL units increase in tumor SUL from the baseline scan in pattern typical of tumor and not of infection/treatment effect or new 18F-FDG avid lesions typical of cancer and not related to treatment effect and/or infection
Arm/Group | Response Evaluation Criteria In Solid Tumors Criteria (RECIST) | PET Response Criteria in Solid Tumours (PERCIST)
Number analyzed (Participants) | 61 | 61
Participants
  Partial response; Partial metabolic response | 5 | 28
  Stable disease; Stable metabolic disease | 41 | 24
  Progressive disease; Progressive metabolic disease | 15 | 9

2. Primary Outcome: Assessment of Early Response by Using 3'-Deoxy-3'-18F-fluorothymidine (18F-FLT) Positron Emission Tomography/Computed Tomography (PET/CT) on Day 21 of Regorafenib Compared With the Response Rate of CT RECIST at 8 Weeks
Description: PET response of 18F-FLT was assessed using the SUVmax. The percentage of change of SUVmax in the target lesion was calculated as follows: 100 ×(SUVmax day 21-SUVmax baseline)/SUVmax baseline. The non responders on 18F-FLT PET/CT were defined as those with decreased SUVmax <10.6% or new lesions on a follow-up scan.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) by CT scans at 8 weeks.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Responders and Non-responders on CT and 18F-FLT PET/CT: By CT scan Responders met the criteria PR according to RECIST criteria. Other than, Non-responders.
  By 18F-FLT PET/CT The non-responders on 18F-FLT PET/CT were defined as those with decreased SUVmax <10.6% or new lesions on a follow-up scan.
  The responders on 18F-FLT PET/CT were defined as those with decreased SUVmax ≥10.6%.
Arm/Group | Responders and Non-responders on CT and 18F-FLT PET/CT
Number analyzed (Participants) | 61
Participants
  Responders on 18F-FLT PET/CT and Responders on RECIST | 5
  Responders on 18F-FLT PET/CT and Non-Responders on RECIST | 43
  Non-Responders on 18F-FLT PET/CT and Responders on RECIST | 0
  Non-Responders on 18F-FLT PET/CT and Non-Responders on RECIST | 13

3. Primary Outcome: Survival Outcomes According to 18F-FLT and 18F-FDG PET/CT Response on Day 21 of Regorafenib and RECIST on CT at 8 Weeks of Regorafenib
Time Frame: Regardless of the reason for discontinuation, all subjects will be followed for survival until death is documented, except for those who specifically withdraw consent to follow-up.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Partial Metabolic Response Group (PMR Group): PMR, Response assessment using 18F-FDG PET/CT was based on the PERCIST 1.0.
- Non-Partial Metabolic Response Group(Non-PMR Group): SMD+PMD, Response assessment using 18F-FDG PET/CT was based on the PERCIST 1.0.
- Non-progressive Metabolic Disease Group (Non-PMD Group): PMR+SMD, Response assessment using 18F-FDG PET/CT was based on the PERCIST 1.0.
- Progressive Metabolic Disease Group (PMD Group): PMD, Response assessment using 18F-FDG PET/CT was based on the PERCIST 1.0.
- Responders on 18F-FLT PET/CT: patients showing a decrease of SUVmax ≥10.6%
- Non-Responders on 18F-FLT PET/CT: patients showing a decrease of SUVmax <10.6% or new lesion.
- Concordant Pairs of Responders on Day 21 18F-FLT PET/CT and 8 Weeks CT: All the responders on 18F-FLT PET/CT met the criteria for responders on 8weeks CT
- Concordant Pairs of Non-responders on Day 21 18F-FLT PET/CT and 8 Weeks CT: All the non-responders on 18F-FLT PET/CT met the criteria for non-responders on 8weeks CT
- Partial Response Group (PR Group): PR, according to RECIST on CT at 8 weeks of Regorafenib.
- Non-Partial Response Group (Non-PR Group): SD+PD, according to RECIST on CT at 8 weeks of Regorafenib.
- Non-Progressive Disease Group (Non-PD Group): PR+SD, according to RECIST on CT at 8 weeks of Regorafenib
- Progressive Disease Group (PD Group): PD, according to RECIST on CT at 8 weeks of Regorafenib
Arm/Group | Partial Metabolic Response Group (PMR Group) | Non-Partial Metabolic Response Group(Non-PMR Group) | Non-progressive Metabolic Disease Group (Non-PMD Group) | Progressive Metabolic Disease Group (PMD Group) | Responders on 18F-FLT PET/CT | Non-Responders on 18F-FLT PET/CT | Concordant Pairs of Responders on Day 21 18F-FLT PET/CT and 8 Weeks CT | Concordant Pairs of Non-responders on Day 21 18F-FLT PET/CT and 8 Weeks CT | Partial Response Group (PR Group) | Non-Partial Response Group (Non-PR Group) | Non-Progressive Disease Group (Non-PD Group) | Progressive Disease Group (PD Group)
Number analyzed (Participants) | 28 | 33 | 52 | 9 | 48 | 13 | 5 | 13 | 5 | 56 | 46 | 15
months
  Progression-free survival(PFS) | 3.9 [1.60 to 6.27] | 3.5 [3.26 to 3.76] | 1.8 [0.00 to 3.79] | 3.6 [3.18 to 4.02] | 3.9 [1.93 to 5.87] | 3.4 [2.72 to 4.16] | 9.0 [2.44 to 15.53] | 3.4 [2.72 to 4.16] | 8.9 [2.43 to 15.53] | 3.5 [3.45 to 3.63] | 5.3 [3.36 to 7.33] | 1.6 [1.33 to 1.88]
  Overall survival (OS) | 11.8 [7.54 to 16.13] | 7.9 [5.25 to 10.62] | 3.9 [2.22 to 6.18] | 10.5 [8.07 to 12.83] | 11.6 [7.33 to 13.85] | 7.0 [4.45 to 9.45] | 10.6 [7.33 to 13.85] | 7.0 [4.45 to 9.45] | 22.5 [0.00 to 45.64] | 9.2 [7.47 to 11.01] | 10.7 [8.00 to 13.37] | 4.6 [1.83 to 7.48]

ADVERSE EVENTS:
Arm/Group | Regorafenib and FLT-PET
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 3/68
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib and FLT-PET (N=68)
hand foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
elevated AST/ALT (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No